CLINICAL TRIAL: NCT05318859
Title: The Safety Assessment of Pharmacopuncture on Musculoskeletal Patients: a Multi-center, Registry
Brief Title: The Safety of Pharmacopuncture on Musculoskeletal Patients
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Hospital director, Research director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2021-17
Record Dates: First submitted 2022-02-11; First posted 2022-04-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Diseases or Conditions; Spine; Arthrosis
Keywords: Spinal joint; Safety; Pharmacopuncture; Adverse Event
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pharmacopuncture — Registry (observational study)

SUMMARY:
The purpose of this study is to evaluate the safety of pharmacopuncture by observing any adverse events that may occur after pharmacopuncture treatment in with spinal joint disease hospitalized patients at 7 Korean medicine hospitals and analyzing blood test results.

DETAILED DESCRIPTION:
This study was an registry observational study, and was conducted in 7 Korean medicine hospitals (160 patients at Jaseng Korean medicine Hospital, 140 patients at Daejeon Jaseng Hospital of Korean Medicine, 140 patients at Bucheon Jaseng Hospital of Korean Medicine, 140 patients at Haeundae Jaseng Korean medicine Hospital, 140 patients at Kyunghee University of Korean medicine Hospital, 140 patients at Kyung Hee University of Korean Medicine Hospital at Gangdong, and 140 patients at Dongguk University Bundang Oriental Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with diagnosed spinal joint disease
* Patients who received pharmacopuncture treatment during hospitalization
* Patients who are 19 years of age or older and less than 70 years old
* Patients who agreed to participate in the clinical study and voluntarily given written informed consent

Exclusion Criteria:

* Patients with difficulty or refusal to give sign written informed consent
* Patients for whom the researchers judge participation in the clinical study to be difficult

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with diagnosed spinal joint disease who are admitted or scheduled to be admitted to Jaseng Hospital of Korean Medicine, Bucheon Jaseng Hospital of Korean Medicine, Daejeon Jaseng Hospital of Korean Medicine, or Haeundae Jaseng Hospital of Korean Medicine, Kyung Hee University Korean Medicine Hospital at Gangdong, Kyung Hee University Korean Medicine Hospital, Dongguk Traditional Herbal Medicine Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of infection cases | 1 month
  Infection is one of the representative adverse events for subcutaneous and intramuscular interventions. Infection cases will be collected to evaluate the safety of pharmacopuncture.

SECONDARY OUTCOMES:
Adverse events | during admission (from day 2 to until discharge), 1 month
  Adverse events refers to undesirable and unintended signs (eg, abnormalities in laboratory test values), symptoms, or diseases that appear after a procedure in the course of a clinical study. Any reported adverse events will be collected to evaluate the safety of pharmacopuncture.
Number of abnormal cases that appeared on the blood analysis | Day 2, discharge day, 1 month
  Any blood analysis result including liver function and renal function will be measured at admission day and discharge moment. The researcher records every abnormal result cases that appeared on the blood analysis and number of abnormal cases will be counted, to evaluate the safety of pharmacopuncture.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Ph.D., Study Director — Jaseng Medical Foundation
Locations (7):
- South Korea (7):
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon, Daejeon
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Kyung Hee University Korean Medicine Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Dongguk University Bundang Oriental Hospital, Seoul